CLINICAL TRIAL: NCT01070004
Title: Countermeasures for Sleepiness at the Wheel and Prediction of Inter- Individual Differences to Their Responses (KillSleep)
Brief Title: Effect of Countermeasures on Nocturnal Driving Performance
Acronym: KILLSLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: ERANET (Unknown); INSERM ERI27 Mobilités Cognition et Temporalité (Unknown); Hotel Dieu Hospital (Other); IMF, CNRS UMR-5231 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2009/14
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Sleepiness
Keywords: sleepiness; driving; countermeasures; coffee; blue light exposure; physical activity
MeSH Terms: conditions — Sleepiness; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blue light (Experimental): Exposure to 460-nm monochromatic light (blue light)
  Interventions: Other: Real driving situation
- Physical activity (Experimental): 15 minutes of physical activity at a low intensity
  Interventions: Other: Driving simulator

INTERVENTIONS:
Other: Real driving situation — Continuous blue light exposure during driving compared to effects of coffee (2*200 mg of caffeine) and coffee placebo on 4h night-time real driving situation. Inside this arm, each volunteer will be randomly allocated and will all receive : continuous blue light exposure, coffee and coffee placebo at each driving session with at least 1 week between each condition.
  Arms: Blue light
Other: Driving simulator — 15 minutes of physical activity at a low intensity before driving compared to effects of coffee (2*200 mg of caffeine) and coffee placebo on 4h night-time driving simulator. Inside this arm, each volunteer will be randomly allocated and will all receive : 15 minutes of physical activity, coffee and coffee placebo at each driving session with at least 1 week between each condition.
  Arms: Physical activity

SUMMARY:
Sleep deprivation induces degradation of night-time driving ability via sleepiness. Because of conflicts between physiological needs and social or professional activities, it is necessary to develop affordable countermeasure to sleepiness. In real-life driving studies, nap and coffee are efficient countermeasures of sleepiness at the wheel. However the effect of caffeine is quick but brief and varies between individuals. There is a need for more knowledge in order to know what to recommend to drivers. Exposure to 460-nm monochromatic light (blue light) decreases subjective sleepiness and improves performances. One objective of this project is to investigate whether blue light exposure during driving would be useful in a real driving situation when sleepiness becomes acute. Owing to the fact that our knowledge of the effects of exercise on driving is very sparse and to the absolutely need to standardize the bouts of exercise that will be applied to the subjects. One objective of the present study will be to investigate in a simulator study the effects of a bout of moderate exercise on participants driving ability when sleepiness becomes acute. Nocturnal neurobehavioral performance varies widely between individuals and only certain subjects seem significantly affected by sleep loss. It is of interest to find biological markers for sleep drive to identify vulnerable drivers to sleep deprivation or to identify responders to sleepiness countermeasures (i.e., coffee and blue light). One objective of this study is to determine individual differences (genetic, hormonal and cognitive) in the impairment of driving skills induced by sleep loss and in the efficiency of countermeasures (blue light and coffee).

ELIGIBILITY:
Inclusion Criteria:

* 20-25-year-old healthy Volunteers or of 40-50 years, male, Caucasian,
* Presenting no disorder of the perception,
* Taking no treatment interfering with the sleep, the attentiveness and the circadian system,
* BMI ≥18 et ≤ 27
* Moderate Drinker of coffee(café) (2-3 cups a day) •
* Presenting no medical history or evolutionary pathology,
* Not presenting syndrome of apneas / hypopnea during the sleep (IAH < 5 for 20-25 years and 10 for 40-50 years),
* Not presenting syndrome of periodic movements during the sleep (Index of MPS < 15),
* Not professional Driver, having their driving license for at least 3 years or 2 years for the drivers who followed the learning anticipated and driving between 10000 and 20000 km a year,
* Having looked in writing their consent to participate in the study,
* Having regular schedules of life 3 days before going into the study,
* Registers on the Social Security and on the register of the healthy volunteers.

Exclusion Criteria:

* Night workers,
* Any evolutionary psychiatric affections (psychosis, disorder(confusion) of the mood or the anxiety),
* All the sleeping disorders (sleep apneas, periodic leg movements, narcolepsy, phase delay, advance of phase),
* Any evolutionary neurological affections (brain tumour, epilepsy, Headache, brain vascular accident, calcifies, myoclonia , chorea, neuropathy, muscular dystrophies, myotonic dystrophy),
* Cardiovascular Pathologies (arterial high blood pressure, cardiac insufficiency, coronary disease, vascular disorders(confusions)),
* Lung Pathologies (BPCO, BPR),
* Renal Disorders(Confusions) (renal insufficiency, nephrolithiases),
* Endocrine Pathologies (dysthyroid, diabetes),
* Drug addiction, alcoholic dependence during the last 6 months,
* Having made a trans-meridian journey (± 3 hours) in last 3 months.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number of inappropriate line crossings identified from video recordings | First, second and third visit

SECONDARY OUTCOMES:
Standard deviation of the position of the car identified from the video recordings | First, second and third visit
Self-rated sleepiness during driving | First, second and third visit
Self-rated fatigue during driving | First, second and third visit
Sleep latency during subsequent sleep | after each driving session
sleep efficiency during the subsequent sleep | after each driving session
Time course of EEG slow wave activity during subsequent sleep | First, second and third visit
Saliva cortisol and amylase concentration | before and after the driving session and after sleep recuperation
Caffeine sensitivity | at first visit
Reaction time and percentage of errors at cognitive tests | First visit
PER3, COMT, ADORA2A and ADA polymorphism | before driving session
Habitual sleep patterns | at first visit
Chronotype | at first visit

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Philip, Pr, Study Director — University Hospital, Bordeaux; Pierre Denise, Pr, Principal Investigator — INSERM ERI27
Locations (2):
- France (2):
  - CHU de Bordeaux Groupe Hospitalier Pellegrin, Bordeaux
  - Université de Caen Basse Normandie, Caen

REFERENCES:
- [Derived] Taillard J, Capelli A, Sagaspe P, Anund A, Akerstedt T, Philip P. In-car nocturnal blue light exposure improves motorway driving: a randomized controlled trial. PLoS One. 2012;7(10):e46750. doi: 10.1371/journal.pone.0046750. Epub 2012 Oct 19. PMID 23094031